CLINICAL TRIAL: NCT02819921
Title: Desvenlafaxine for the Treatment of Hot Flashes in Women With Breast Cancer Taking Tamoxifen: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Desvenlafaxine for Treatment of Hot Flashes in Women With Breast Cancer Taking Tamoxifen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in Recruiting Research Participants
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Korea Cancer Center Hospital (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WI209149
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hot Flashes; Breast Neoplasms
Keywords: Hot Flashes; Breast Neoplasms; Tamoxifen; Desvenlafaxine Succinate
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Desvenlafaxine succinate 100mg (Experimental): Titration with 50 mg Desvenlafaxine succinate tablet once daily for 1 week, then 2 tablets of 50mg Desvenlafaxine succinate tablet once daily for 3 weeks, then taper with 50 mg Desvenlafaxine succinate tablet once daily for 3 days.
  Interventions: Drug: Desvenlafaxine succinate 100mg
- Desvenlafaxine succinate 50mg (Experimental): 50 mg Desvenlafaxine succinate tablet once daily for 1 week, then 1 tablets of 50mg Desvenlafaxine succinate tablet and 1 tablet of 50mg placebo tablet once daily for 3 weeks, then 50mg placebo tablet once daily for 3 days.
  Interventions: Drug: Desvenlafaxine succinate 50mg
- Placebo (Placebo Comparator): 50 mg placebo tablet once daily for 1 week, then 2 tablets of 50mg placebo tablet once daily for 3 weeks, then 50 mg placebo tablet once daily for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine succinate 100mg — Pristiq 100mg
  Arms: Desvenlafaxine succinate 100mg
Drug: Desvenlafaxine succinate 50mg — Pristiq 50mg
  Arms: Desvenlafaxine succinate 50mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled study of desvenlafaxine versus placebo. The purpose of this study is to determine if desvenlafaxine was effective in decreasing the frequency and severity of hot flashes in breast cancer patients taking tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

i. Women age 18 years and older with localized breast cancer. Histologic documentation of atypical ductal hyperplasia, ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), or invasive adenocarcinoma of the breast stages I-III A.

ii. Current daily tamoxifen use (≥ 6 days/week). Any planned surgery, adjuvant chemotherapy or radiation must have been completed.

iii. History of bothersome hot flushes: ≥ 14 hot flushes/week (average ≥ 2 hot flushes/day), sufficiently severe that intervention is desired. Participants must have had bothersome hot flushes for at least one month prior to enrollment.

Exclusion Criteria:

i. Women who is pregnant or breast feeding, or who has a history of seizure disorder or hepatic or renal insufficiency ii. Concurrent systemic hormone replacement therapy (estrogen, progestational agents, androgens) or use of corticosteroids iii. Concurrent use of other antidepressants, anxiolytics and antipsychotics, gabapentin, pregabalin and clonidine for treatment of hot flushes or depression.

iv. Presense or past history of severe psychiatric symptoms such as hallucinations and delusions, manic episodes, or high suicide risk.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Reduction rate of hot flashes symptom score | From baseline to Week 5 (Intervention is started from Week 1)
  Participants would complete self -report daily diary on which they record the number and severities (1 - 4 points) of hot flashes from baseline to week 5. Each symptom severities are multiplied by the numbers of symptoms to determine the daily hot flashes symptom score. The mean of daily hot flashes symptom score of one week is calculated and regared as a hot flashes symptom score for the week. The efficacy of Desvenlafaxine is assessed by comparing the reduction rate of weekly hot flashes symptom score (= hot flashes symptom score at week 5 - hot flashes symptom score at baseline / hot flashes symptom score of baseline) for each group.

SECONDARY OUTCOMES:
Clinical impression state and change | Week 1, Week 2, Week 5
  Clinical global impression (CGI) would be used to assess clinical impression state and change.
Peripheral neuropathy | Week 1, Week 2, Week 5
  European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy(EORTC-QLQ-CIPN-20) would be used to assess peripheral neuropathy.
Depression | Baseline, Week 2, Week 5
  Patient health questionnaire (PHQ-9) would be used to assess mood status.
Anxiety | Baseline, Week 2, Week 5
  Generalized anxiety disorder-7 (GAD-7) would be used to assess anxiety.
Manic or Hypomanic symptoms. | Baseline, Week 2, Week 5
  Mood disorder questionnaire (MDQ) would be used to assess manic or hypomanic symptoms.
Sleep quality | Baseline, Week 2, Week 5
  Pittsburgh sleep quality index (PSQI) would be used to assess sleep quality.
Chonotype | Baseline
  Morningness-Eveningness questionnaire (MEQ) would be used to assess chronotype.
Circadian misalignment | Baseline, Week 2, Week 5
  Munich Chronotype Questionnaire (MCTQ) would be used to assess circadian misalignment.
Fatigue | Baseline, Week 2, Week 5
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-fatigue) would be used to assess fatigue.
Quality of life | Baseline, Week 2, Week 5
  Functional Assessment of Cancer Therapy-Breast (FACT-B) would be used to assess quality of life.
Beliefs about medicines | Baseline
  Beliefs about Medicines Questionnaire (BMQ) would be used to assess beliefs about medicines.
Illness perception | Baseline
  Brief Illness Perception Questionnaire (BIPQ) would be used to assess illness perception.
Social support | Baseline
  Multidimensional Scale of Perceived Social Support (MSPSS) would be used to assess social supports.
Body image | Baseline
  Body Image Scale (BIS) would be used to assess body image.
Resilience | Baseline
  Connor-Davidson Resilience Scale (CDRS) would be used to assess resilience.
Hormonal level | Week 2
  Serum estradiol, follicle-stimulating hormone (FSH) and anti-Müllerian hormone (AMH) levels would be used to examine pathophysiological mechanisms associated with the presence of hot flashes, mood status and desvenlafaxine treatment.
Genetic polymorphism | Week 2
  estrogen receptors (ESR1 PvuII; rs#2234693 and XbaI; rs#9340799 and ESR2-02; rs#4986938) and serotonin transporter gene (SLC6A4; rs#11080121) would be used to examine pathophysiological mechanisms associated with the presence of hot flashes, mood status and desvenlafaxine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Jin Hahm, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim Y, Yeom CW, Lee HJ, Kim JH, Lee KM, Kim TY, Lee HB, Kim H, Im SA, Lee KH, Kim M, Han W, Moon HG, Spiegel D, Hahm BJ, Son KL. Differential effects of desvenlafaxine on hot flashes in women with breast cancer taking tamoxifen: a randomized controlled trial. NPJ Breast Cancer. 2024 Jul 17;10(1):59. doi: 10.1038/s41523-024-00668-w. PMID 39019875